CLINICAL TRIAL: NCT04049318
Title: Effects of a Structured Digital Osteoarthritis Self-management Program After 6 Months of Adherence
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: X
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Exercise; Education; Digital treatment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 24 weeks: Subjects who participated in the intervention who have data available at week 24
  Interventions: Other: Education+ exercise (delivered digitally)
- 48 weeks: Subjects who participated in the intervention who have data available at week 48
  Interventions: Other: Education+ exercise (delivered digitally)

INTERVENTIONS:
Other: Education+ exercise (delivered digitally) — The intervention consisted of a digital, structured and individualized treatment program for people with hip or knee OA (Joint Academy®; www.jointacademy.com). The program consists of neuromuscular exercises appropriately adjusted to each patient in regard to degrees of complexity and difficulty, continuous access to and dialogue with a physiotherapist through a chat function, and/or telephone , and information in the form of text or video lessons (with quizzes on the material after each episode) on subjects related to OA, OA symptoms and its management.

SUMMARY:
This is a study based on a cohort in a register of patients enrolled in a digital osteoarthritis self-management program, Joint Academy. The purpose of this study is to examine joint pain and the potential change of this pain, in patients with long-term adherence to a digital self-management program for individuals with knee- and hip osteoarthritis. The hypothesis, based on preliminary findings is that pain levels of those adhering to the program, decreases over time. To test the hypothesis, participants weekly pain report will be investigated whilst adhering to the digital program for 6- to 12 months, and statistically tests will be performed to find out whether significant differences can be seen over time.

DETAILED DESCRIPTION:
Introduction Osteoarthritis (OA) is highly prevalent in older adults and a growing cause of disability. The importance of availability of primary treatment of OA is gaining momentum, and web-based self-management programs have in recent years become available. Evidence of short term effects of such programs are abundant, yet the evaluation of long term effects of these programs is scarce.

Aim To investigate joint pain development over time from participation in a web-based OA self-management program for people with hip or knee OA.

Methods Participants joined the program through advertisements and campaigns on the web. Included participants had a radiographic or clinical diagnosis of hip or knee OA (about 95%) from a physical therapist or physician. The intervention consisted of a digital, structured and individualized treatment program for people with hip or knee OA (Joint Academy®; www.jointacademy.com). The program consists of neuromuscular exercises appropriately adjusted to each patient in regard to degrees of complexity and difficulty and information in the form of text or video lessons (with quizzes on the material after each episode) on subjects related to OA, OA symptoms and its management.

Outcome measures Joint pain in the hip or knee was assessed at baseline, and weeks 12, 24 and 48 using the Numerical Rating Scale (NRS), a 0-10 scale where 0 is defined as No pain and 10 is defined as Maximum pain. Minimal clinically important change (MCIC) of pain was defined as an improvement of 20%. As a measure of physical function, the 30-second chair stand test (30CST) was used and performed by the patient every other week, using an instruction video with a coupled visual timer. The patient entered the performed number of repetitions after each test. Physical function data was handled similarly to the NRS, with week 24 ±4 adjacent weeks and week 48±6 adjacent weeks included for those with available NRS data. All outcomes were self-assessed, self-centred, and chosen based on the International Consortium for Health Outcomes Measurement Standard Set for Hip & Knee Osteoarthritis (ICHOM).

Statistical analysis Summary data are described by the mean value, standard deviation and number of observations or the number and percent of the categories of interest. The group-specific mean treatment effect of duration on pain and repetitions (30CST - physical function), as well as differences in pain over time between hip and knee OA with or without additional covariates, were estimated and tested using random slopes and intercepts models. Pain development over time was plotted for hip and knee OA respectively.

To describe patients adhering for six months with contrasting pain severity at baseline, participants were divided into same-sized tertiles based on reported baseline pain, with related descriptive data. Mean pain per time point was calculated and plotted for each group. Significance level was set to p<0.05, and p-values and 95% confidence intervals were reported when applicable. Statistical calculations were performed in Statistical Package for Social Sciences (SPSS Version 25, IBM Corporation, New York, USA) and Stata 15.1 (StataCorp LLC, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* radiographic or clinical diagnosis of hip or knee OA (about 95%) from a physical therapist or physician
* had been treated in the digital non-surgical treatment program the first 3 weeks with a adherence of at least 70%
* had been included in the program at least 24 weeks prior to the data extraction

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: At the time of the study start (13th of March, 2019), the Joint Academy patient database contained data from 1709 Swedish participants who had reported one of their knees or hips as their most symptomatic joint
Sampling Method: Non-Probability Sample
Enrollment: 1709 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Change in NRS pain | 0-24 and 0-48 weeks
  0 no pain, 10 max pain
Change in 30 second chair stand test (30CST) | 0-24 and 0-48 weeks
  sit to stand repetitions in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Nero, PhD, Principal Investigator — Lund University
Locations (1):
- Arthro therapeutics, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorstensson CA, Garellick G, Rystedt H, Dahlberg LE. Better Management of Patients with Osteoarthritis: Development and Nationwide Implementation of an Evidence-Based Supported Osteoarthritis Self-Management Programme. Musculoskeletal Care. 2015 Jun;13(2):67-75. doi: 10.1002/msc.1085. Epub 2014 Oct 24. PMID 25345913
- [Background] Cronstrom A, Dahlberg LE, Nero H, Ericson J, Hammarlund CS. 'I would never have done it if it hadn't been digital': a qualitative study on patients' experiences of a digital management programme for hip and knee osteoarthritis in Sweden. BMJ Open. 2019 May 24;9(5):e028388. doi: 10.1136/bmjopen-2018-028388. PMID 31129601
- [Background] Nero H, Ranstam J, Kiadaliri AA, Dahlberg LE. Evaluation of a digital platform for osteoarthritis treatment: study protocol for a randomised clinical study. BMJ Open. 2018 Nov 8;8(11):e022925. doi: 10.1136/bmjopen-2018-022925. PMID 30413507
- [Background] Nero H, Dahlberg J, Dahlberg LE. A 6-Week Web-Based Osteoarthritis Treatment Program: Observational Quasi-Experimental Study. J Med Internet Res. 2017 Dec 18;19(12):e422. doi: 10.2196/jmir.9255. PMID 29254906
- [Background] Cronstrom A, Nero H, Dahlberg LE. Factors Associated With Patients' Willingness to Consider Joint Surgery After Completion of a Digital Osteoarthritis Treatment Program: A Prospective Cohort Study. Arthritis Care Res (Hoboken). 2019 Sep;71(9):1194-1201. doi: 10.1002/acr.23772. Epub 2019 Jul 17. PMID 30298990